CLINICAL TRIAL: NCT03436498
Title: Safety Assessment of SAR341402 and NovoLog® Used in Continuous Subcutaneous Insulin Infusion (CSII) in Adult Patients With Type 1 Diabetes Mellitus (T1DM)
Brief Title: Safety Assessment of SAR341402 and NovoLog® Used in Continuous Subcutaneous Insulin Infusion for Type 1 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PDY15083; U1111-1200-1241 (Other: UTN)
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR341402/NovoLog (Experimental): SAR341402 will be self-administered via continuous subcutaneous insulin infusion via an insulin pump. The dose will be individually titrated and administered in a basal and bolus fashion. After 4 weeks of SAR341402 as treatment, patient will switch with NovoLog® as treatment.
  Interventions: Drug: Insulin aspart SAR341402
- NovoLog/SAR341402 (Experimental): Novolog will be self-administered via continuous subcutaneous insulin infusion via an insulin pump. The dose will be individually titrated and administered in a basal and bolus fashion. After 4 weeks of NovoLog® as treatment, patient will switch with SAR341402 as treatment.
  Interventions: Drug: Insulin aspart

INTERVENTIONS:
Drug: Insulin aspart SAR341402 — Pharmaceutical form: Solution
  Route of administration: Subcutaneous
  Arms: SAR341402/NovoLog
Drug: Insulin aspart — Pharmaceutical form: Solution
  Route of administration: Subcutaneous
  Arms: NovoLog/SAR341402

SUMMARY:
Primary Objective:

- To assess the safety of SAR341402 and NovoLog® when used in external insulin pumps in terms of the number of patients with infusion set occlusions.

Secondary Objectives:

* To assess the safety of SAR341402 and NovoLog® when used in external pumps in terms of unexplained hyperglycemia.
* To assess the safety of SAR341402 and NovoLog® when used in external pumps in terms of:
* Intervals for infusion set changes.
* Number of patients with insulin pump for "non-delivery" alarm.
* Patient observation of infusion set occlusion.
* Adverse events and serious adverse events.
* Number of patients with hypoglycemic events [according to ADA (American Diabetes Association) Workgroup on hypoglycemia].

DETAILED DESCRIPTION:
The study duration for each patient will be approximately 10 weeks, including a 2-week screening period, 2 treatment periods of 4 weeks each, and 1-day post-treatment safety follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients with Type 1 diabetes mellitus (T1DM).
* Age greater than or equal to 18 at the screening visit.
* Diabetes diagnosed at least 12 months before screening visit.
* At least 1 year of insulin treatment with at least 6 months of CSII (Continuous Subcutaneous Insulin Infusion) treatment with an external insulin pump.
* Demonstration of successful use of insulin pump and performing of a minimum of 4 blood glucose checks per day during screening.
* Laboratory parameters within the normal range (or defined screening threshold for the Investigator site), unless the Investigator considers an abnormality to be clinically irrelevant for T1DM patients.
* Signed written informed consent.

Exclusion criteria:

* Hemoglobin A1c (HbA1c) ≥8.5% at screening.
* Diabetes other than T1DM.
* History of infection at the infusion site within 3 months prior to the screening visit (Visit 1).
* Use of oral glucose-lowering agents or any injectable glucose-lowering agents other than insulin during the 3 months before screening visit.
* Hospitalization for recurrent diabetic ketoacidosis (DKA) in the last 6 months before screening visit.
* History of severe hypoglycemia requiring emergency room admission or hospitalization in the last 6 months before screening visit.
* Hypoglycemic unawareness as judged by the Investigator in the last 6 months before the screening visit.
* Any clinically significant abnormality identified on physical examination, laboratory tests, or vital signs at the time of screening that in the judgment of the investigator or any sub investigator would preclude safe completion of the study.
* Known history of illegal drug or alcohol abuse within 6 months prior to the time of screening.
* Use of investigational drug(s) within 3 months or 5 half-lives, whichever is longer, prior to the screening visit.
* Patients who had previously received SAR341402 in any other clinical trial.
* Any contraindication to the use of NovoLog® as defined in the national product labels; history of hypersensitivity to NovoLog® or to any of the excipients.
* Pregnancy and lactation.
* If female, pregnancy [defined as positive β-HCG (Human Chorionic Gonadotropin) in blood or in urine], breast-feeding.
* Patient is an employee or relative of an employee of the sponsor.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2018-10-06 (Actual); Study Completion 2018-10-06 (Actual)

PRIMARY OUTCOMES:
Infusion set occlusions | At week 4 from baseline of each treatment
  Number of patients with infusion set occlusions. Infusions set occlusions are defined as infusion set change due to failure to correct hyperglycemia (plasma glucose ≥ 250 mg/dL [13.9 mmol/L]) by insulin bolus via the insulin pump.

SECONDARY OUTCOMES:
Unexplained hyperglycemia | At week 4 from baseline of each treatment
  Number of patients with unexplained hyperglycemia. Unexplained hyperglycemia is defined as plasma glucose equal or above 250 mg/dL (13.9 mmol/L) whether or not corrected by a bolus through the insulin pump with no apparent material defects, medical, dietary, insulin dosing or pump failure. This will include infusion set occlusion as defined in the primary endpoint.
Intervals for infusion set changes | At week 4 from baseline of each treatment
  Intervals for infusion set changes will be derived as number of days in the treatment period divided by the number of infusion set changes in the treatment period.
Number of patients with insulin pump alarms for "non-delivery" | At week 4 from baseline of each treatment
  Number of patients with insulin pump "non-delivery" alarms (independent of confirmation of occlusion by hyperglycemia and failure to correct hyperglycemia by insulin bolus via the insulin pump).
Patient observation of infusion set occlusion | Up to 10 weeks
  Patient observation of infusion set occlusion (independent of confirmation of occlusion by hyperglycemia and failure to correct hyperglycemia by insulin bolus via the insulin pump).
Adverse events and serious adverse events | Up to 10 weeks
  Number patients with adverse events and/or serious adverse events, including bruising at the infusion site and injection site, and hypersensitivity reactions.
Number of patients with hypoglycemic events | At week 4 from baseline of each treatment
  Number of patients with hypoglycemic events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Investigational Site Number 8400001, Little Rock, Arkansas
  - Investigational Site Number 8400002, Denver, Colorado
  - Investigational Site Number 8400003, West Des Moines, Iowa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Thrasher J, Polsky S, Hovsepian L, Nowotny I, Pierre S, Bois De Fer B, Bhargava A, Mukherjee B, Garg SK. Safety and Tolerability of Insulin Aspart Biosimilar SAR341402 Versus Originator Insulin Aspart (NovoLog) When Used in Insulin Pumps in Adults with Type 1 Diabetes: A Randomized, Open-Label Clinical Trial. Diabetes Technol Ther. 2020 Sep;22(9):666-673. doi: 10.1089/dia.2019.0446. Epub 2020 Jan 28. PMID 31833801